CLINICAL TRIAL: NCT00720785
Title: Safety and the Anti- Tumor Effects of Escalating Doses of Adoptively Infused Ex Vivo Expanded Autologous Natural Killer (NK) Cells Against Metastatic Cancers or Hematological Malignancies Sensitized to NK-TRAIL Cytotoxicity With Bortezomib
Brief Title: Natural Killer Cells and Bortezomib to Treat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080186; 08-H-0186
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-07-14

CONDITIONS: Chronic Myeloid Leukemia (CML); Pancreatic Ca; Colon/Rectal Ca; Multiple Myeloma; Carcinoma, Non-Small -Cell Lung
Keywords: Metastatic Solid Tumor; Chronic Myelogenous Leukemia (CML); Small Lymphocytic Lymphoma (SLL); Chronic Lymphocytic Leukemia (CLL); Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): NK Cell Infusion (cell /kg pt wt)
  Interventions: Biological: NK cells
- 2 (Experimental): 1.3 mg/m2/dose administered as a 3 to 5 second bolusintravenous injection
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Parenteral formulation. It is supplied as a 3.5 mg single use vial containing a sterile lyophilized powder that requires reconstitution.
  Arms: 2
Biological: NK cells — NK Cell Infusion
  Arms: 1

SUMMARY:
Natural killer (NK) cells are white blood cells that have a limited ability to kill cancer cells. This ability might be enhanced if they are given 24 hours after an injection of the drug bortezomib. This study will determine the following:

* What dose of NK cells can be given safely to subjects with metastatic solid tumors or leukemia.
* The effectiveness and side effects of NK cell therapy
* How the body handles NK cells.

People between 18 and 70 years of age who have a solid tumor or leukemia, and for whom standard treatments are not effective, may be eligible for this study. Participants undergo the following procedures:

Apheresis to collect NK cells. For this procedure, a catheter (plastic tube) is placed in a vein in the subject s arm. Blood flows from the vein into a cell separator machine, which separates the white cells from the other blood components. The white cells are extracted and the rest of the blood is returned to the body through a second tube placed in a vein in the other arm.

Chemotherapy with the drug pentostatin to suppress the immune system and prevent it from attacking the NK cells that will be infused.

Chemotherapy with bortezomib to increase NK cell function.

Infusion of the NK cells. In this dose-escalating study, successive groups of patients entering the study receive increasingly higher numbers of cells to determine the highest safe dose level. Up to ten dose levels may be studied.

Interleukin-2 drug therapy to maintain NK cell activity.

Evaluations during therapy including:

* Clinical assessment, history and review of medications
* Blood draws for routine and research tests.
* Pharmacokinetics study after the NK infusion to see how the body handles the cells. For this test, the number of NK cells in the blood are measured over time. This requires drawing about 1 teaspoon of blood at 15 minutes, 30 minutes, 1, 2, 4, 8, 12, and 24 hours after the infusion (day 1); then every 24 hours on days 2 through 7, then once on days 10, 14, and 21.
* Bone marrow biopsy (subjects with leukemia only).
* Chest x-ray.
* CT scan, bone scan and PET scan, if indicated, for disease evaluation.

Subjects who respond well after one treatment cycle may be eligible to continue NK cell therapy.

...

DETAILED DESCRIPTION:
Natural killer (NK) cells are innate immune lymphocytes that are identified by the expression of the CD56 surface antigen and the lack of CD3. Unlike antigen specific T cells, NK cells do not require the presence of a specific tumor antigen for the recognition and killing of cancer cells. Our in vitro studies have demonstrated that pretreatment of malignant cells with bortezomib significantly enhances NK-mediated tumor cytotoxicity by sensitizing cells to TNF-related apoptosis-inducing ligand (TRAIL). TRAIL is a member of tumor necrosis factor family of cytokines that promotes apoptosis. Importantly, in our laboratory, in vitro expanded NK cells isolated from patients with metastatic cancers or hematological malignancies exhibited significantly more cytotoxicity against their tumor cells when tumors were pre-treated with bortezomib compared with untreated tumor controls. These findings suggest that drug-induced sensitization to TRAIL could be used as a novel strategy to potentiate anticancer effects of autologous adoptively infused NK cells in patients with cancer.

Murine studies conducted in our laboratory have also established that bortezomib treatment sensitizes tumors in vivo to killing by adoptively infused syngeneic NK cells; murine renal cell carcinoma line (RENCA) tumors in BALB/c mice grew significantly slower and survival was prolonged when syngeneic NK cell infusions where given following bortezomib treatment compared to mice receiving NK cell infusions alone or bortezomib alone. This anti-tumor effect was further potentiated by eradicating T-regulatory cells prior to adoptive NK cell infusion and by administering interleukin-2 after adoptive NK cell infusion.

Recently, our laboratory has developed techniques for the in vitro isolation and expansion of NK cells to levels suitable for the treatment of cancer patients. Furthermore, we have also established good viability and sterility of these expanded NK cells which, compared to fresh NK cells, have increased surface expression of TRAIL and have enhanced cytotoxicity against tumor cells.

We therefore propose this non-randomized, Phase I, dose escalating study designed to evaluate the safety and the anti- tumor effects of escalating doses of adoptively infused ex vivo expanded autologous natural killer (NK) cells against metastatic cancers or hematological malignancies sensitized to NK TRAIL cytotoxicity with bortezomib.

The primary study objective is to determine the safety (maximum tolerated dose) of escalating NK cell doses of adoptively infused ex vivo expanded autologous NK cells in subjects with treatment refractory metastatic tumors or hematological malignancies that are sensitized to NK cell cytotoxicity using bortezomib. Secondary objectives will include the anti-neoplastic effects of this treatment regimen (assessed using standard disease specific response criteria) and the toxicity profile associated with extended cycles of protocol therapy.

The primary endpoint will be assessed at day 21 (3 weeks after the Day 0 NK cell infusion).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosed with histologically confirmed metastatic solid tumor - cancer of the lung (small cell or non small cell), prostate (adenocarcinoma), colorectum, kidney (renal cell carcinoma), pancreas (adenocarcinoma),or malignant melanoma, metastatic Ewing's sarcoma, or metastatic epithelial neoplasms and adenocarcinoma of unknown primary, and disease confirmed to be metastatic and unresectable for which standard curative or beneficial treatments are no longer effective

     OR

     Diagnosed with a hematological malignancy (multiple myeloma, [MM] chronic myelogenous leukemia [CML] or chronic lymphocytic leukemia [CLL] or small lymphocytic lymphoma [SLL]) and disease resistant or refractory to standard therapy and CLL/SLL patients are required to have failed prior treatment with at least one nucleoside analogue. Myeloma patients are required to have disease which has progressed following treatment with bortezomib.
  2. At least 4 weeks since any prior systemic therapy (excluding corticosteroid therapy) to treat the underlying malignancy (standard or investigational). NOTE: subjects on FDA-approved tyrosine kinase inhibitors or other targeted therapies for RCC such as mTOR inhibitors that have evidence of disease progression on therapy may continue these medicines until the time of study enrollment (as accelerated disease progression following discontinuation of these drugs has been described).
  3. At least 2 weeks since prior palliative radiotherapy.
  4. Ages greater than or equal to 18 years and less than or equal to 70 years.
  5. Evidence of progressive disease over a 3-month interval.
  6. RBC transfusion independent (solid tumor patients only).

EXCLUSION CRITERIA:

1. Disease not evaluable radiographically (applies to solid tumor patients only).
2. Disease involving greater than 25% of the liver radiographically (estimated based on review of liver lesions seen on CT scan).
3. History of an allogeneic hematopoietic stem cell transplant.
4. Brain metastases (with the exception of patients with a single brain metastasis less than 1cm treated with either sterotactic or gamma knife radiotherapy) due to poor prognosis and potential for neurological dysfunction that would confound evaluation of neurological and other adverse events).
5. Peripheral neuropathy of grade greater than 1, which would require reduction of bortezomib dose.
6. Acute diffuse infiltrative pulmonary disease.
7. Acute pericardial disease.
8. Life expectancy less than 3 months.
9. ECOG performance status 2, 3 or 4.
10. Uncontrolled concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, life threatening cardiac arrhythmia. Patients with symptoms of coronary artery disease, cardiac arrhythmias or an abnormal thallium stress test must be evaluated and cleared by cardiology prior to enrollment.
11. Ongoing or active infection
12. Contraindication for administration of pentostatin, bortezomib, and/or interleukin-2.
13. Allergy or hypersensitivity to bortezomib, boron or mannitol by history.
14. Concurrent use of corticosteroids.
15. For all tumor types:

    Marrow function characterized by

    -Absolute neutrophil count less than 500/mcL (must be present off growth factors)

    Organ function characterized by
    * Total bilirubin greater than 3 times upper limit of normal
    * AST (SGOT)/ALT (SGPT) greater than 4 times upper limit of normal
    * Creatinine clearance less than 50 cc/min based on a 24 hour urine collection
    * Left ventricular ejection fraction less than 40% by echocardiogram (ECHO)
    * Hypercalcemia greater than 2.5 mmol/L

    For all Hematologic malignancies:

    Marrow function characterized by
    * Neutrophil count less than or equal to 500/mcl
    * Platelets less than or equal to 20,000/mcl
16. HIV-positive patients
17. Hepatitis C positive patients (Hep C PCR positive)
18. Active Hepatitis B infection (Hep B surface antigen positive)
19. Pregnant or nursing
20. Psychiatric illness/social situations that would limit compliance with study requirements and ability to comprehend the investigational nature of the study and provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
safety of escalating NK cell doses of adoptively infused ex vivo expanded autologous NK cells in subjects with treatment refractory metastatic tumors or hematological malignancies that are sensitized to NK cell toxicity with bortezomib. | After each 3 week cycle
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Last J. Informed consent/consentement eclaire. Ann R Coll Physicians Surg Can. 1992 Aug;25(5):263-4. No abstract available. PMID 11651409
- [Background] Farag SS, Caligiuri MA. Human natural killer cell development and biology. Blood Rev. 2006 May;20(3):123-37. doi: 10.1016/j.blre.2005.10.001. Epub 2005 Dec 20. PMID 16364519
- [Background] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- [Background] Gautier JF, Ravussin Y. A New Symptom of COVID-19: Loss of Taste and Smell. Obesity (Silver Spring). 2020 May;28(5):848. doi: 10.1002/oby.22809. Epub 2020 Apr 1. No abstract available. PMID 32237199
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-H-0186.html